CLINICAL TRIAL: NCT04660227
Title: Effectiveness of Exercise Training in Pediatric-Onset Multiple Sclerosis Patients
Brief Title: Exercise Training in Pediatric-Onset Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Pelin Vural, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IU-C2020-26
Record Dates: First submitted 2020-11-25; First posted 2020-12-09 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Pediatric Multiple Sclerosis
Keywords: Physical Activity; Physiotherapy; Degenerative diseases; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Participants in the online exercise program group will be given a treatment protocol consisting of aerobic exercise and strengthening exercises in the presence of a physiotherapist for a total of 8 weeks, 2 days a week for 1 hour.
  Interventions: Procedure: Exercise Trainning
- Control Group (Other): Participants in the control group will be put on the waiting list after all assessment methods have been applied and will be re-evaluated at the end of 8 weeks.
  Interventions: Other: Control Group

INTERVENTIONS:
Procedure: Exercise Trainning — Participants in the online exercise program group will be given a treatment protocol consisting of aerobic exercise and strengthening exercises in the presence of a physiotherapist for a total of 8 weeks, 2 days a week for 1 hour. Before starting the exercise, the risk of possible injury will be minimized by doing warm-up exercises and preparations will be made to start the exercise. Then, the exercise program will be started with aerobic exercise. Strengthening exercises will be planned for large muscle groups, targeting body parts such as hips, knees, shoulders, abdomen and trunk. In exercises, it is planned to do 2 sets of 10-15 repetitions using elastic band, free weights or body weight. The exercise program will be created according to the condition of the people and progression will be provided every 2 weeks. After the exercises are completed, cool down will be done with relaxation and stretching exercises.
  Arms: Exercise Group
Other: Control Group — Participants in the control group will be put on the waiting list after all assessment methods have been applied and will be re-evaluated at the end of 8 weeks. After the final evaluations, they will be directed to the exercise group.
  Arms: Control Group

SUMMARY:
Multiple sclerosis is one of the leading causes of disability in young adults. It is known that patients with pediatric onset multiple sclerosis (POMS) experience their first demyelinating attack before the age of 18. However, studies conducted with individuals with pediatric onset of multiple sclerosis have been reported to be few and have affected parameters such as physical activity, fatigue balance and quality of life. Therefore, this study is planned to consist of two stages. These are the following stages;

1. Assessment of people with pediatric onset multiple sclerosis with the evaluation methods detailed below. After these evaluations, the relationship between the 6-minute walk test performance of the patients and other evaluations will be examined. Within the scope of the project, a publication will be prepared and uploaded with the data obtained from this stage.
2. The patients are divided into two groups, one group is included in the online exercise program, and the other group is included in the exercise program after being put on the waiting list.

DETAILED DESCRIPTION:
People with pediatric onset multiple sclerosis (POMS) experience various sensory, motor, cerebellar and cognitive dysfunctions due to the destruction of the central nervous system. These disorders may cause limitation of physical activity in people with POMS. In a study comparing people with POMS with monophasic acquired demyelinating syndrome (mono-ADS) and healthy controls in terms of physical activity levels, it was reported that people with POMS performed less physical activity compared to other groups. In addition, it has been reported that people with POMS have increased complaints such as depression and fatigue and their quality of life decreases. The aim of this study is to (1) investigate functional exercise capacity and its relationship between physical activity level, muscle strength, balance, fatigue and quality of life in POMS patients and (2) examine the effect of online exercise training on physical activity, balance, fatigue and quality of life in POMS patients. Participants will be randomly divided into two groups, the online exercise program group and the control group, after the evaluations. Participants in the online exercise program group will be given a treatment protocol consisting of aerobic exercise and strengthening exercises in the presence of a physiotherapist for a total of 8 weeks, 1 hour on 2 days a week. The exercise program will be created according to the condition of the people and progression will be provided every 2 weeks. After the exercises are completed, cooling will be done with stretching exercises. Participants in the control group will be put on the waiting list after all assessment methods are applied and will be re-evaluated at the end of 8 weeks. Application of the exercise training online will prevent the difficulties of continuing the exercise program due to transportation problems, disability level or pandemic and will facilitate the participation of people with POMS in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with pediatric onset multiple sclerosis
* EDSS <6
* Having internet access

Exclusion Criteria:

* Having an orthopedic problem affecting its mobility
* Blurred vision problem
* Having another diagnosis in addition to the diagnosis of pediatric onset multiple sclerosis
* Having had an attack or received corticosteroid treatment 3 months before participating in the study

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
The Leisure-Time Exercise Questionnaire (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a self-reported questionnaire with two questions that measures the physical activity behavior of the participants. In the first question, the frequencies of mild, moderate and intense physical activity performed for more than 15 minutes in a normal week are questioned. Weekly frequencies of light, moderate, and vigorous physical activities are multiplied by 3, 5 and 9 metabolic equivalents, respectively, and the sum of the results is recorded as total leisure activity. Second question seeks the frequency of activity that causes sweating in a normal week is questioned. Less than 14 scores means insufficiently active/sedentary, 14-23 scores means moderately active and 24 scores or more means active. So higher scores better outcomes.
One-Week Step Count Measurement with Pedometer for Physical Activity Assessment (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is one of the objective methods used to evaluate physical activity. It is used to record the number of steps taken. The estimated step length is entered into the device and recorded as a step when the vertical oscillation of the body exceeds a certain threshold value. In our study, the number of steps taken by the participants during a week before and after treatment will be calculated and recorded. Higher scores better outcomes.

SECONDARY OUTCOMES:
Evaluation of Isokinetic Muscle Strength of Quadriceps and Hamstring Muscles with Biodex Multi-Joint System (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  Evaluation of muscle strength will be made with "Biodex Multi-Joint System" isokinetic device. Isokinetic tests are evaluations that allow the measurement of muscle strength, strength and endurance with an isokinetic device at constant angular velocity and constant resistance objectively. Angular velocities to be used during the test are between low 30-60°/s , medium 90-120°/s and high 180-300°/s. Force tests are performed at low speeds, and strength and endurance tests are performed at high speeds. In our study, the concentric isokinetic muscle strength of the knee flexor and extensor muscles for the lower extremity at angular speeds of 30, 60 and 90°/s will be evaluated.
Knee Joint Proprioception Assessment with Biodex Multi-Joint System (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  Participants' knee joint proprioception will be evaluated using the Biodex Multi-Joint System. To show the participant the target angles, the participant's leg will be passively moved to the target angles and the knee will be held in the target position for 10 seconds and then brought back to the starting position (90°). The participant will then be asked to bring the index to the chosen target angle and press the stop button when bringing the index to the target angle. Each test attempt will be performed three times after a 30-second rest in a quiet environment. An eye patch will be used to prevent the use of visual inputs during the test. By measuring the target position three times, the average joint position absolute error degrees will be calculated. A lower mean absolute error value indicates better knee proprioception.
Static and Dynamic Postural Stability Assessment with Biodex Balance System (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  The Biodex Balance System is a platform that allows an objective assessment of the participant's ability to regulate his balance while standing on a stable or unstable surface. In our study, the postural stability abilities of the participants will be evaluated. The assessment will measure the General Stability Index, anterior/posterior stability index and medial/lateral stability index. Each participant will be asked to take a postural stance on the balance platform with bare feet, with eyes open and as still as possible for 20 seconds. Postural stability assessment in Biodex Balance System is applied on two different grounds as static and dynamic ground. While the static evaluation surface is fixed, the dynamic evaluation will be tested at the stability level 7 of the surface. Evaluation results will be recorded with the automatic reporting of the Biodex Balance System at the end of the evaluation.
6 Minute Walk Test (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a simple, practical test applied according to the standard protocol of the American Thoracic Society to measure walking capacity. It has been reported that the test is valid and reliable in MS patients with mild and moderate disability. In our study, 6 MWTs will be performed in accordance with the standards set in the guidelines for MS patients. The participant will be asked to walk as fast as possible at his own walking pace on the 30-meter track for 6 minutes. Before starting the test, participants will be explained that they can rest if they develop excessive fatigue or respiratory distress during the test and that this time is included in the test period. As a result of the test, the distance traveled by the participant will be recorded in meters.
Timed 25-Foot Walk (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a performance test that provides information about the participant's mobility and leg function. The standardized protocol is very simple. The participant will be requested to walk as quickly and safely as possible (ie maximum walking speed) along a clearly marked, linear 25 feet or 7.62 m track. The participant can use an assistive device while walking. The person will walk two different times on the marked track and the average of two consecutive attempts in seconds will be recorded as a result of the test.
Timed Up and Go (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a test used to evaluate dynamic balance. The test measures the time it takes a participant to get up from the chair and walk 3 meters at a comfortable pace and return to the chair and sit down. The test begins when the participant gets up from the chair and ends when the participant sits down on the chair again. The time measured is recorded in seconds. A shorter period represents better mobility.
The Pediatric Quality of Life Inventory 4.0 (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  The Pediatric Quality of Life Inventory is a 23-item multidimensional inventory that includes: 1- Physical Functions (8 Items), 2- Emotional Functions (5 Items), 3- Social Functions (5 Items), and 4- School Functions (5 Items). The inventory includes two parallel forms, the Child and Family form. In the inventory prepared according to the five-point Likert system, questions are scored between 0-4 points. In calculating the total score of the scale, a linear transformation is applied and an evaluation is made over 0-100 points. Therefore, the higher the Pediatric Quality of Life Inventory score indicates that the health-related quality of life is better.
Fatigue Severity Scale (The change between the initial value and the value after 2 months will be evaluated). | Baseline and end of weeks 8.
  It is a scale that evaluates the fatigue of MS patients in daily functions. In the evaluation made with 9 questions, each question is scored between 1 (totally disagree) - 7 (totally agree). The result score is the average value of nine questions. High score indicates increased severity of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Vural, Principal Investigator — Istanbul University-Cerrahpasa Institute of Postgraduate Education; Yonca Zenginler Yazgan, PhD, Study Chair — Istanbul University-Cerrahpasa Faculty of Health Science; Sema Saltık, Prof. Dr., Study Chair — Istanbul University-Cerrahpasa Cerrahpasa Faculty of Medicine, Department of Pediatric Neurology; Serhat Güler, Assoc. Prof., Study Chair — Istanbul University-Cerrahpasa Cerrahpasa Faculty of Medicine Department of Pediatric Neurology
Locations (1):
- Istanbul University-Cerrahpasa, Bakırköy, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Grover SA, Aubert-Broche B, Fetco D, Collins DL, Arnold DL, Finlayson M, Banwell BL, Motl RW, Yeh EA. Lower physical activity is associated with higher disease burden in pediatric multiple sclerosis. Neurology. 2015 Nov 10;85(19):1663-9. doi: 10.1212/WNL.0000000000001939. Epub 2015 Aug 12. PMID 26268901
- [Background] Grover SA, Sawicki CP, Kinnett-Hopkins D, Finlayson M, Schneiderman JE, Banwell B, Till C, Motl RW, Yeh EA. Physical Activity and Its Correlates in Youth with Multiple Sclerosis. J Pediatr. 2016 Dec;179:197-203.e2. doi: 10.1016/j.jpeds.2016.08.104. Epub 2016 Oct 4. PMID 27717498
- [Background] Sikes EM, Richardson EV, Motl RW. A Qualitative Study of Exercise and Physical Activity in Adolescents with Pediatric-Onset Multiple Sclerosis. Int J MS Care. 2019 Mar-Apr;21(2):81-91. doi: 10.7224/1537-2073.2018-033. PMID 31049039
- [Background] Storm Van's Gravesande K, Blaschek A, Calabrese P, Rostasy K, Huppke P, Kessler J J, Kalbe E, Mall V; MUSICADO Study group. Fatigue and depression predict health-related quality of life in patients with pediatric-onset multiple sclerosis. Mult Scler Relat Disord. 2019 Nov;36:101368. doi: 10.1016/j.msard.2019.08.010. Epub 2019 Aug 9. PMID 31557681
- [Background] Hebert D, Geisthardt C, Hoffman H. Insights and Recommendations From Parents Receiving a Diagnosis of Pediatric Multiple Sclerosis for Their Child. J Child Neurol. 2019 Jul;34(8):464-471. doi: 10.1177/0883073819842420. Epub 2019 Apr 23. PMID 31012369
- [Background] Weikert M, Motl RW, Suh Y, McAuley E, Wynn D. Accelerometry in persons with multiple sclerosis: measurement of physical activity or walking mobility? J Neurol Sci. 2010 Mar 15;290(1-2):6-11. doi: 10.1016/j.jns.2009.12.021. Epub 2010 Jan 8. PMID 20060544
- [Background] Warren JM, Ekelund U, Besson H, Mezzani A, Geladas N, Vanhees L; Experts Panel. Assessment of physical activity - a review of methodologies with reference to epidemiological research: a report of the exercise physiology section of the European Association of Cardiovascular Prevention and Rehabilitation. Eur J Cardiovasc Prev Rehabil. 2010 Apr;17(2):127-39. doi: 10.1097/HJR.0b013e32832ed875. PMID 20215971
- [Background] Moghadasi A, Ghasemi G, Sadeghi-Demneh E, Etemadifar M. The Effect of Total Body Resistance Exercise on Mobility, Proprioception, and Muscle Strength of the Knee in People With Multiple Sclerosis. J Sport Rehabil. 2020 Feb 1;29(2):192-199. doi: 10.1123/jsr.2018-0303. PMID 30676232
- [Background] Abdin MMN, Abdelazeim F, Elshennawy S. Immediate effect of induced fatigue of the unaffected limb on standing balance, proprioception and vestibular symptoms in children with hemiplegia. J Pediatr Rehabil Med. 2020;13(2):119-125. doi: 10.3233/PRM-180587. PMID 32444572
- [Background] Greve JM, Cug M, Dulgeroglu D, Brech GC, Alonso AC. Relationship between anthropometric factors, gender, and balance under unstable conditions in young adults. Biomed Res Int. 2013;2013:850424. doi: 10.1155/2013/850424. Epub 2013 Jan 16. PMID 23509788
- [Background] Soysal Tomruk M, Uz MZ, Kara B, Idiman E. Effects of Pilates exercises on sensory interaction, postural control and fatigue in patients with multiple sclerosis. Mult Scler Relat Disord. 2016 May;7:70-3. doi: 10.1016/j.msard.2016.03.008. Epub 2016 Mar 22. PMID 27237762
- [Background] Paltamaa J, West H, Sarasoja T, Wikstrom J, Malkia E. Reliability of physical functioning measures in ambulatory subjects with MS. Physiother Res Int. 2005;10(2):93-109. doi: 10.1002/pri.30. PMID 16146327
- [Background] Marrie RA, Goldman M. Validity of performance scales for disability assessment in multiple sclerosis. Mult Scler. 2007 Nov;13(9):1176-82. doi: 10.1177/1352458507078388. Epub 2007 Jul 10. PMID 17623733
- [Background] Rampello A, Franceschini M, Piepoli M, Antenucci R, Lenti G, Olivieri D, Chetta A. Effect of aerobic training on walking capacity and maximal exercise tolerance in patients with multiple sclerosis: a randomized crossover controlled study. Phys Ther. 2007 May;87(5):545-55. doi: 10.2522/ptj.20060085. Epub 2007 Apr 3. PMID 17405806
- [Background] Savci S, Inal-Ince D, Arikan H, Guclu-Gunduz A, Cetisli-Korkmaz N, Armutlu K, Karabudak R. Six-minute walk distance as a measure of functional exercise capacity in multiple sclerosis. Disabil Rehabil. 2005 Nov 30;27(22):1365-71. doi: 10.1080/09638280500164479. PMID 16372431
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Motl RW, Cohen JA, Benedict R, Phillips G, LaRocca N, Hudson LD, Rudick R; Multiple Sclerosis Outcome Assessments Consortium. Validity of the timed 25-foot walk as an ambulatory performance outcome measure for multiple sclerosis. Mult Scler. 2017 Apr;23(5):704-710. doi: 10.1177/1352458517690823. Epub 2017 Feb 16. PMID 28206828
- [Background] Sönmez, S., & Başbakkal, Z. (2007). Türk Çocuklarının Pediatrik Yaşam Kalitesi 4. Envanterinin (PedsQL 4.) Geçerlilik ve Güvenilirlik Çalışması. Türkiye Klinikleri Pediatri Dergisi, 16(4), 229-237.
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071